CLINICAL TRIAL: NCT05685160
Title: Ultrasound and MRI of the Forefoot: Intermetatarsal Bursitis or Morton's Neuroma
Brief Title: US and MRI of the Forefoot: Intermetatarsal Bursitis or Morton's Neuroma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Danish Rheumatism Association (Other); Hvidovre University Hospital (Other); Bispebjerg Hospital (Other); Gentofte Hospital (Unknown)
Responsible Party: Principal Investigator, Sif Binder Larsen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-20067346
Record Dates: First submitted 2022-12-06; First posted 2023-01-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Intermetatarsal Bursitis; Morton Neuroma; Intermetatarsal Neuroma
Keywords: Forefoot pain; Metatarsalgia
MeSH Terms: conditions — Morton Neuroma; Metatarsalgia | interventions — Magnetic Resonance Imaging; Ultrasonography

STUDY DESIGN:
Intervention Model Description: This is a diagnostic study with a patient and a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient group (Experimental): Patients with intermetatarsal pain have ultrasound and MRI done
  Interventions: Diagnostic Test: MRI with contrast; Diagnostic Test: Ultrasound
- Control group (Active Comparator): Healthy individuals (no forefoot pain) undergo ultrasound and MRI scan of the forefoot.
  Interventions: Diagnostic Test: MRI with contrast; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: MRI with contrast — MRI of the forefoot with contrast (Gadovist)
Diagnostic Test: Ultrasound — Ultrasound imaging of the forefoot

SUMMARY:
The aim of this study is to investigate the incidence of intermetatarsal bursitis and Morton's neuroma in patients with metatarsalgia (i.e. pain in the forefoot) and control subjects by diagnostic imaging with ultrasound and MRI.

DETAILED DESCRIPTION:
In a group of patients with intermetatarsal pain found by an orthopedic surgeon, the investigators want to assess the incidences of intermetatarsal bursitis and Morton's neuroma, using diagnostic imaging; ultrasound and MRI.

The hypothesis is, that intermetatarsal bursitis is an overlooked diagnosis in patients with metatarsalgia. As a result of sparse literature and lack of knowledge about this condition with symptoms mimicking Morton's neuroma, a part of patients diagnosed with Morton's neuroma, suffers from intermetatarsal bursitis instead.

Additionally, the investigators want to evaluate the clinical sign opening toes.

Based on clinical photos of the feet, the investigators want to document the presence of opening toes and investigate if there is a correlation with either intermetatarsal bursitis and/or Morton's neuroma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Pain in an intermetatarsal space (patient group)

Exclusion Criteria:

* Age <18 years
* Open wounds or ongoing infection in the forefoot at the time of examination
* Persons with contraindications to participate in MRI scan
* Persons with a history of significant trauma in the forefoot, e.g. any fracture or previous surgeries in the forefoot
* Persons who have previously received treatment for Morton's neuroma in the same foot, e.g. injection (within 6 months) or operation (anytime)
* Persons with severely impaired renal function (GFR <30 ml/min)
* Persons with a systemic inflammatory condition like rheumatoid arthritis, due to clinically silent intermetatarsal bursitis in this group (control group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of intermetatarsal bursitis on MRI | 8 weeks
  High intensity on T2 weighted images, low signal on T1. Thin peripheral enhancement on T1 contrast enhanced pictures.
Incidence of intermetatarsal bursitis on US | 8 weeks
  Hypoechoic mass between metatarsal heads closest to dorsal surface of foot. Compressible. Activity on power/color doppler.
Incidence of Morton's neuroma on MRI | 8 weeks
  Low to Intermediate signal in T1 and T2. Contrast enhancement of the nodular focus.
Incidence of Morton's neuroma on US | 8 weeks
  Hypoechoic mass between metatarsal heads closest to plantar surface of foot. Non-compressible. The interdigital nerve can be seen entering the mass. Close relation to the interdigital artery.
Incidence of other pathology on MRI | 8 weeks
  Other pathology than intermetatarsal bursitis or Morton's neuroma.
Incidence of other pathology on US | 8 weeks
  Other pathology than intermetatarsal bursitis or Morton's neuroma.
Incidence of normal findings on MRI | 8 weeks
  When no findings is observed.
Incidence of normal findings on US | 8 weeks
  When no findings is observed.

SECONDARY OUTCOMES:
Opening toes | 8 weeks
  Presence of opening toes/V-sign/spreading toes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Copenhagen, Denmark